CLINICAL TRIAL: NCT04377412
Title: Risk Factors for Anxiety and Depression Among Pregnant Women During the COVID-19 Pandemic - a Web-based Cross-sectional Survey
Brief Title: Risk Factors for Anxiety and Depression Among Pregnant Women During the COVID-19 Pandemic
Acronym: MindCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Żelazna Medical Centre, LLC (Other)
Collaborators: University of Medicine, Tirana (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Charles University, Czech Republic (Other); Hôpital Necker-Enfants Malades (Other); Charite University, Berlin, Germany (Other); Chinese University of Hong Kong (Other); Meir Medical Center (Other); Università degli Studi di Brescia (Other); American University of Beirut Medical Center (Other); Karolinska Institutet (Other); Pomeranian Medical University Szczecin (Other); Nicolaus Copernicus University (Other); Centre of Postgraduate Medical Education (Other); Polish Academy of Sciences (Other); Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other); Fundación Para la Investigación y el Desarrollode la Medicina Materno-Fetal y Neonatal "iMaterna", Madrid (Unknown); Taiji Clinic, Taipei (Unknown); Wayne State University (Other); Chang Gung University (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Anna Kajdy, Md, PhD, Centre of Postgraduate Medical Education
Other Study IDs: Maternal axiety and COVID-19
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Depression; Pregnancy Related
Keywords: coronavirus; mental health; pregnancy; anxiety; depression; COVID-19; pandemic
MeSH Terms: conditions — Anxiety Disorders; Depression; Coronavirus Infections; Psychological Well-Being; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Albania
  Interventions: Other: Pandemic control measures
- Australia
  Interventions: Other: Pandemic control measures
- Czech Republic
  Interventions: Other: Pandemic control measures
- France
  Interventions: Other: Pandemic control measures
- Germany
  Interventions: Other: Pandemic control measures
- Hong Kong
  Interventions: Other: Pandemic control measures
- Israel
  Interventions: Other: Pandemic control measures
- Italy
  Interventions: Other: Pandemic control measures
- Lebanon
  Interventions: Other: Pandemic control measures
- Norway
  Interventions: Other: Pandemic control measures
- Poland
  Interventions: Other: Pandemic control measures
- Russia
  Interventions: Other: Pandemic control measures
- Spain
  Interventions: Other: Pandemic control measures
- Sweden
  Interventions: Other: Pandemic control measures
- Taiwan
  Interventions: Other: Pandemic control measures
- Ukraine
  Interventions: Other: Pandemic control measures
- United States
  Interventions: Other: Pandemic control measures

INTERVENTIONS:
Other: Pandemic control measures — Population of different countries are exposed to different pandemic control measures, and everyday lives of pregnant women are affected on different levels. Investigators will measure influence their influence on mental health.

SUMMARY:
The article presents a protocol of a cross-sectional study of mental health of pregnant women in relation to the COVID 19 pandemic. The primary aim is to compare differences in anxiety and depression scores of pregnant women between countries affected by the COVID-19 pandemic. The secondary aim is to assess demographic, economic, and social aspects affecting maternal anxiety and depression scores among pregnant women worldwide in the time of the COVID-19 pandemic. Finally, investigators will be able to compare differences in perception of the different aspects of the COVID-19 pandemic (social distancing, restrictions related to delivery) between countries and according to the epidemic status (number of infected patients, number of reported deaths). The comparisons will also be done according to COVID-19 status of the participants.

ELIGIBILITY:
Inclusion Criteria:

* declaration of being pregnant
* being able to complete the survey in the available languages
* answer the screening questions
* provide informed consent for participation

Exclusion Criteria:

* not providing online informed consent for participation
* if the participant does not click on the submit button at the end of the survey
* not answer all the GAD-7 and PHQ-9 scale questions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: About 10% of pregnant women experience perinatal depression globally. Untreated perinatal depression may result in adverse obstetric outcomes and is a risk factor for poor maternal health, inadequate prenatal care, and postpartum depression. In addition to the potential negative impact on pregnancy outcomes, perinatal depression is associated with disrupted maternal-infant bonding, increased irritability, and decreased activity. Children born to depressed mothers are at risk for delayed cognitive and language development, lower IQ, and increased prevalence of psychiatric and emotional problems. Depression that begins during pregnancy frequently continues or worsens after delivery.
Sampling Method: Non-Probability Sample
Enrollment: 8500 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 4 months
  Anxiety measured by General Anxiety Disorder-7 (GAD-7) scale. Scoring:5-9 mild; 10-14 moderate; >15 severe. Minimum 0, maximum 21 points
Depression | 4 months
  Depression measured by Patient Health Questionnaire-9 (PHQ-9) scale. Scoring: 5-9 mild;10-14 moderate; 15-19 moderately severe; >20 severe. Minimum 0 maximum 27 points

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kajdy, MD, PhD, Study Chair — Centre of Postgraduate Medical Education; Michał Rabijewski, MD, PhD, Professor, Principal Investigator — Centre of Postgraduate Medical Education; Dorota Sys, PhD, Principal Investigator — Centre of Postgraduate Medical Education; Jan Modzelewski, MD, Principal Investigator — Centre of Postgraduate Medical Education; Sebastian Kwiatkowski, MD, PhD, Principal Investigator — Pomeranian Medical University Szczecin; Roksana Lewandowska, MD, Principal Investigator — Pomeranian Medical University Szczecin; Dariusz Borowski, MD, PhD, Principal Investigator — Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz; Barbara Baranowska, PhD, RM, Principal Investigator — Centre of Postgraduate Medical Education; Artur Pokropek, PhD, Professor, Principal Investigator — Institute of Philosophy and Sociology of the Polish Academy of Sciences; Urszula Ajdacka, MD, Principal Investigator — Central Clinical Hospital of Ministry of Internal Affairs and Administration; Stepan Feduniw, MD, Principal Investigator — Żelazna Medical Centre; Medical Faculty od Lazarski University; Maria del Mar Gil Mira, MD, PhD, Principal Investigator — Fundación Para la Investigación y el Desarrollode la Medicina Materno-Fetal y Neonatal "iMaterna"; Simone Schwank, PhD M.S. M.A. Msc. Clinical Ps, Principal Investigator — Karolinska Institutet; Ksenia Olisova, MD, MPH, Principal Investigator — Taiji Clinic, Taipei; Tung-Yao Chang, MD, M Med Sci, Principal Investigator — Taiji Clinic, Taipei; Steven Shaw, Principal Investigator — Chang Gung University; Sonia Hassan, MD, Principal Investigator — Wayne State University; Jade Harris, MD, Principal Investigator — Wayne State University; Orion Gliozheni, MD, Principal Investigator — University of Medicine, Tirana; Jon Hayett, Professor, Principal Investigator — Royal Prince Alfred Hospital, Sydney; Pavel Calda, MD, MSc, Professor, Principal Investigator — Charles University, Czech Republic; Laurent J Salomon, MD, PhD, Professor, Principal Investigator — Université de Paris; Stefan Verlohren, MD, Professor, Principal Investigator — Charite University, Berlin, Germany; Liona C Poon, MBBS, MRCOG, Professor, Principal Investigator — Chinese University of Hong Kong; Tal Biron-Shental, MD, Principal Investigator — Meir Medical Center; Maya Ben-Zion, MD, Principal Investigator — Meir Medical Center; Federico Prefumo, MD, PhD, Principal Investigator — Università degli Studi di Brescia; Gihad Chalouhi, MD, PhD, Principal Investigator — American University of Beirut Medical Center; Ganesh Acharya, MD, PhD, FRCOG, Professor, Principal Investigator — Karolinska Institutet; Heidi Tiller, MD, PhD, Principal Investigator — The Arctic University of Norway; Karine Stiberg Birkelund, Principal Investigator — The Arctic University of Norway; Solrun Rasmussen, Principal Investigator — The Arctic University of Norway; Ewa Andersson, RNM, PhD, Principal Investigator — Karolinska Institutet
Locations (17):
- Wayne State University, Detroit, Michigan, United States
- University of Medicine Tirana, Tirana, Albania
- Royal Prince Alfred Hospital, Sydney, Australia
- Charles University, Prague, Czechia
- Université de Paris, Paris, France
- Charité - University Medicine Berlin, Berlin, Germany
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Meir Medical Center, Kafr Saba, Israel
- University of Brescia, Brescia, Italy
- American University of Beirut, Beirut, Lebanon
- The Arctic University of Norway, Tromsø, Norway
- Poland (3):
  - Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz, Bydgoszcz
  - Pomeranian Medical University, Szczecin
  - Centre of Postgraduate Medical Education, Warsaw
- 11. Fundación Para la Investigación y el Desarrollode la Medicina Materno-Fetal y Neonatal "iMaterna", Madrid, Spain
- Karolinska Institutet, Stockholm, Sweden
- Taiji Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided